CLINICAL TRIAL: NCT05154162
Title: Prospective Multi-centre Randomised Trial of the Additive Diagnostic Value of PSMA PET in Men With Negative/Equivocal MRI in the Diagnosis of Significant Prostate Cancer
Brief Title: PSMA PET Additive Value for Prostate Cancer Diagnosis in Men With Negative/Equivocal MRI
Acronym: PRIMARY2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Collaborators: St Vincent's Hospital, Sydney (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20/043
Record Dates: First submitted 2021-10-25; First posted 2021-12-10 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
Keywords: Prostate; Cancer; PSMA PET
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): Pelvic PSMA PET ± transperineal targeted prostate biopsy
  Interventions: Diagnostic Test: PSMA PET/CT; Procedure: Transperineal targeted prostate biopsy
- Control (Other): No pelvic PSMA PET + transperineal template prostate biopsy
  Interventions: Procedure: Transperineal template prostate biopsy

INTERVENTIONS:
Diagnostic Test: PSMA PET/CT — PSMA PET/CT (limited to the pelvis)
  Arms: Experimental
Procedure: Transperineal template prostate biopsy — Transperineal template prostate biopsies will be performed as per treating urologist's usual practice. No specific template for biopsy is prescribed for the purposes of the study. However, template sampling of the prostate is required, with a minimum of 12 cores, dependent on prostate volume. MRI will be available for any additional targeted biopsies required. Transperineal template biopsies must be labelled appropriately and sent for histopathological analysis.
  Arms: Control
Procedure: Transperineal targeted prostate biopsy — If the PSMA PET/CT is normal, transperineal prostate biopsy would be omitted If the PSMA PET/CT is abnormal, transperineal prostate biopsies would be performed targeting the MRI (done prior to study) and PSMA PET/CT images
  Arms: Experimental

SUMMARY:
This clinical trial will evaluate PSMA PET additive value for significant prostate cancer (sPCa) diagnosis in men with negative/equivocal MRI

DETAILED DESCRIPTION:
This open label, phase III, multi-centre, randomised trial with a non-inferiority objective will evaluate the additive diagnostic value of PSMA PET for men with negative/equivocal MRI in the diagnosis of significant prostate cancer. Patients with a clinical suspicion of prostate cancer with PI-RADS 2 or 3 on MRI, meeting all the inclusion and none of the exclusion criteria will be randomised into experimental and control arms. Patients in the experimental arm would be subjected to Pelvic PSMA PET/CT, wherein the PSMA negative patients would not undergo biopsy as opposed to PSMA positive patients who will be subjected to Transperineal targeted prostate biopsy. Whereas patients in the control arm will only receive Standard of Care (SOC) with no additional imaging (PSMA PET) and will undergo Transperineal template prostate biopsy. The co-primary objectives are to assess (1) the percentage of men with sPCa in the experimental arm (transperineal targeted biopsy) compared to the control arm (transperineal template biopsy) defined as the presence of a single biopsy core indicating disease Gleason score (GS) 3+4(>10%)=7, grade group (GG) 2, and (2) the percentage of men who avoid transperineal prostate biopsy between both arms. The secondary objectives include determining the percentage of clinically insignificant PCa on targeted biopsy (experimental arm) versus transperineal template biopsy (control arm); estimating the difference in complications from transperineal prostate biopsy between both arms; the health economics impact between the experimental and control arms; estimating the mean difference between both arms in change from baseline in health-related quality of life (QoL); estimating the mean difference between both arms at each time point in generalised anxiety and cancer worry.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all the following criteria for study entry:

  1. Males aged ≥ 18 years at the time of consent
  2. No previously diagnosed prostate cancer
  3. No previous prostate biopsy
  4. Having undergone MRI within 9 months prior to randomisation and meet one of the following criteria:

     * PI-RADS 2 AND ≥1 red flag defined as:

       * PSA density >0.1
       * Abnormal DRE
       * Strong family history (1 first degree relative or ≥2 second degree)
       * BRCA mutation
       * PSA >10
       * PSA doubling time <36 months
       * PSA velocity >0.75/year
     * PI-RADS 3
  5. Intention for prostate biopsy
  6. Willing and able to comply with all study requirements

Exclusion Criteria:

* Patients who meet any of the following criteria will be excluded from study entry:

  1. Having a PSA >20ng/ml
  2. Having ≥ cT3 on DRE
  3. Significant morbidity that, in the judgement of the investigator, would limit compliance with study protocol

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males aged ≥ 18 years at the time of consent
Enrollment: 660 (Estimated)
Dates: Start 2022-03-02 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Presence of sPCa on prostate biopsy | When histology results are available, at an expected average of 14 days post-biopsy
  sPCa defined as Gleason score 3+4(>10%)=7, Grade group 2 Patients without biopsy (negative PSMA PET) are considered not to have sPCa.
Number of men who avoid transperineal prostate biopsy in the experimental arm | When the PSMA PET result is available, at most 28 days after randomisation
  In the experimental arm, if PSMA PET is negative, the patient does not have biopsy

SECONDARY OUTCOMES:
Presence of insignificant prostate cancer (isPCa) on prostate biopsy | Within 3 months following randomisation
  isPCa defined as GS 3+3=6, GG 1 or GS 3+4(≤10%)=7, GG 2
Cost per quality adjusted life year | Through study completion, estimated up to 2 years
  cost-effectiveness analysis to assess the cost per quality adjusted life year (QALY) gained associated with the use of PSMA PET in addition to MRI compared with MRI alone for the diagnosis of sPCa. Importantly, this analysis will take into consideration the impact on costs and QoL associated with the hypothesised reduction in unnecessary biopsies arising from the improved accuracy of PSMA+MRI and the comparative interventions).
Health-related quality of life as measured by the EORTC QLQ-C30. | Within 7 days of randomisation and every 6 months ± 30 days after randomisation
  Quality of life (QoL) will be assessed using QLQ-C30, which contains 30 items across five functional scales, three symptom scales, global health status, and six single items. Participant responses are collected using a four-point response scale ranging from 'Not at all' to "Very much". Higher scores indicate better QoL and function, while high scores for the symptom scale represent a high level of symptoms.
Anxiety as measured by the GAD7 in the diagnosis of PCa. | Within 7 days following randomisation and every 6 months ± 30 days after randomisation
  The generalized anxiety disorder Scale (GAD-7)14 is a 7-item, patient-rated questionnaire for screening and severity measuring of generalised anxiety disorder. The GAD-7 score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of 'not at all', 'several days', 'more than half the days', and 'nearly every day', respectively, and adding together the scores for the seven questions. Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively.
Cancer worry in the diagnosis of PCa. | Within 7 days following randomisation and every 6 months ± 30 days after randomisation
  The modified Cancer Worry Scale adaptation of Cancer Worry Scale is a 3-item questionnaire used in context of cancer worry in abnormal PSA levels in men participating in community screening program. The score is calculated by assigning scores of 1, 2, 3, and 4, to the categories 'not at all or rarely', 'sometimes', 'often', and 'a lot', respectively, and adding together the scores for the 3 questions. A final question asks about feelings of distress related to cancer risk.
Number of biopsy cores | Within 3 months following randomisation
  Experimental arm: For patients with a positive PSMA PET, the images, the report and a simplified template will be made available to the treating urologist. Up to four identified lesions on PSMA PET and/or MRI will be targeted with each lesion having a minimum 5 cores.
  Control arm: Transperineal template prostate biopsies will be performed as per treating urologist's usual practice. No specific template for biopsy is prescribed for the purposes of the study. However, template sampling of the prostate is required, with a minimum of 12 cores,dependent on prostate volume.
Incidence of complications following transperineal prostate biopsy. | Within 7 days following randomisation and at 3 and 6 months after randomisation
  Complications following biopsy will be assessed with a modified questionnaire validated in the PRECISION trial. Part 1 following randomisation is a 9 item questionnaire. Part 2 is a 23 item questionnaire administered at 3 and 6 months to assess complications from transperineal prostate biopsy. The following complications will be assessed via these forms: fever, blood in urine, blood in semen, blood in stool, acute urinary retention, erectile dysfunction, urinary incontinence, urinary tract infection and pain in the perineum.
Incidence of erectile dysfunction following transperineal prostate biopsy | Within 7 days following randomisation and at 3 and 6 months after randomisation
  The Sexual Health Inventory for Men (SHIM) is an adapted version of the 5 item International Index of Erectile Function (IIEF-5) score, developed to diagnose the presence and severity of erectile dysfunction. This validated questionnaire has a range of scores from 1 to 25, grading erectile dysfunction into 5 categories (none, mild, mild to moderate, moderate and severe).
Number of men who have sPCa detected only with PSMA PET (MRI PI-RADS 2) | Within 28 days following randomisation
  Measured in the experimental arm in patients with positive PSMA PET and negative MRI (PIRADS 2). sPCa defined as Gleason score 3+4(>10%)=7, Grade group 2

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hofman, Principal Investigator — Peter MacCallum Cancer Centre, Australia; Louise Emmett, Principal Investigator — St Vincent's Sydney; Mark Frydenberg, Principal Investigator — Cabrini Health; Sze-Ting Lee, Principal Investigator — Austin Health; Matthew Roberts, Principal Investigator — Royal Brisbane and Women's Hospital; Yang Du, Principal Investigator — Royal Adelaide Hospital
Locations (6):
- Australia (6):
  - St Vincent's Hospital, Sydney, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Austin Health, Melbourne, Victoria
  - Cabrini Health, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Buteau JP, Moon D, Fahey MT, Roberts MJ, Thompson J, Murphy DG, Papa N, Mitchell C, De Abreu Lourenco R, Dhillon HM, Kasivisvanathan V, Francis RJ, Stricker P, Agrawal S, O'Brien J, McVey A, Sharma G, Levy S, Ayati N, Nguyen A, Lee SF, Pattison DA, Sivaratnam D, Frydenberg M, Du Y, Titus J, Lee ST, Ischia J, Jack G, Hofman MS, Emmett L. Clinical Trial Protocol for PRIMARY2: A Multicentre, Phase 3, Randomised Controlled Trial Investigating the Additive Diagnostic Value of [68Ga]Ga-PSMA-11 Positron Emission Tomography/Computed Tomography in Men with Negative or Equivocal Multiparametric Magnetic Resonance Imaging for the Diagnosis of Clinically Significant Prostate Cancer. Eur Urol Oncol. 2024 Jun;7(3):544-552. doi: 10.1016/j.euo.2023.11.008. Epub 2023 Dec 6. PMID 38061976